CLINICAL TRIAL: NCT03415009
Title: Prevalence of IL28B Polymorphism in Hepatitis C Patients in Singapore and Its Effect on the Outcome of Hepatitis C Treatment
Brief Title: Prevalence of IL28B Polymorphism in Hepatitis C Patients
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CG12Aug02-13
Record Dates: First submitted 2016-02-16; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Hepatitis C
Keywords: IL28B gene
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from whole blood sample will be used as template for real-time PCR amplification. It will be analyzed for the genotypes of IL28B SNPs (genotype CC/CT/TT for rs12979860 and TT/GT/GG for rs8099917).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCV genotype 1 and genotype 2/3: DNA extracted from whole blood sample will be used as template for real-time PCR amplification. It will be analyzed for the genotypes of IL28B SNPs (genotype CC/CT/TT for rs12979860 and TT/GT/GG for rs8099917).

SUMMARY:
Response to peginterferon and ribavirin treatment in hepatitis C (HCV) depends on viral and host factors. Single nucleotide polypmorphisms (SNP) near to IL28B gene (especially at rs12979860 and rs8099917) are strongly associated with the response to treatment in HCV genotype 1 infection, less so in HCV genotype 2/3 infection. CC genotype in rs12979860 and TT genotype at rs8099917 are associated with good treatment outcome. Asian populations have high prevalence of CC genotype in other studies, which can explain relatively good response to peginterferon/ ribavirin in genotype 1 infection in Asians compared with Caucasians.

DETAILED DESCRIPTION:
The prevalence of different genotypes of IL28B polymorphism in the local population will be studied. DNA will be extracted from the whole blood sample of hepatitis C patients with genotype 1, 2 and 3 infection. It will be amplified by real-time PCR and subsequently analysed for the genotypes of IL28B SNPs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive HCV IgG (EIA or RIBA test) and positive HCV RNA test (RT-PCR)
* HCV genotypes 1, 2 or 3 (determined by Versant™ HCV genotype Assay LiPA 2.0)
* with or without HCV treatment (peginterferon/ ribavirin).

Exclusion Criteria:

-Patients with acute hepatitis C infection.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatitis C patients with genotype 1, 2/3
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
the prevalence of genetic variants for IL28B SNPs (rs 12979860 and rs 8099917) in HCV patients in Singapore. | Baseline

SECONDARY OUTCOMES:
The distribution of the different SNP variants in different ethnic groups (Chinese, Malay, Indian and others) | Baseline
The association of the genetic variants and the treatment response in patients receiving peg-interferon/ ribavirin therapy. | Baseline
  To study the correlation between genetic variants and treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Poh Yen Loh, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes